CLINICAL TRIAL: NCT06209853
Title: Correlation Between Prostate-Specific Antigen (PSA) Levels and Fluorine-18 Prostate-Specific Membrane Antigen Positron Emission Tomography/Computed Tomography (F-18 PSMA PET/CT) Scan Findings in Patients With Prostate Cancer
Brief Title: Correlation Between PSA Levels and F-18 PSMA PET/CT Findings in Prostate Cancer Patient
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aalaa Wael Hussein, Assistant Lecturer, Assiut University
Other Study IDs: F-18 PSMA in prostate cancer
Record Dates: First submitted 2024-01-06; First posted 2024-01-18 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Prostatic Neoplasms
Keywords: PSMA PET/CT, Prostate, PSA
MeSH Terms: conditions — Prostatic Neoplasms; Salivary Gland Adenoma, Pleomorphic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PSMA PET/CT — Patients need no specific preparation. F-18 PSMA dose will be 3-4 MBq/kg and injected via IV route scan will be performed 90-120 min after injection

SUMMARY:
It is a cross sectional study aimed to correlate between PSA Levels and F-18 PSMA PET/CT Scan findings and to evaluate the impact of PET/CT findings on the patient management

DETAILED DESCRIPTION:
Prostate cancer (PC) is a prevalent malignancy that occurs primarily in old males, it is the third most common with regards of mortality (1,2). prostate-specific membrane antigen (PSMA) known as glutamate carboxypeptidase II, is a transmembrane glycoprotein highly expressed in PC cells. PSMA expression tends to increase with increased pathological Gleason grade and is thought to be upregulated with the emergence of androgen independence (2).

PSMA PET/CT imaging is important for correct primary staging and for the detection of sites of biochemical recurrence.

prostate-specific antigen Liu et al., in 2022 stated that as serum PSA levels increase, the diagnostic accuracy of F-PSMA-1007 PET/CT also improves (3) Bergero et al., in 2022 evaluated the diagnostic correlation between PSA and positivity of F-18 PSMA PET/CT in patients with biochemically recurrent prostate cancer (RPC), reporting it as a very good predictor of positivity in 18F-PSMA PET/CT in patients with RPC (4).

A Meta-Analysis in 2022 found that the detection rate (DR) of the18F-PSMA-1007 PET/CT was also improved with increasing serum PSA levels (5) Another Meta-Analysis in 2019 studied the DR of F-18 PSMA PET/CT revealing that DR is related to PSA values with significant lower DR in patients with PSA<0.5 ng/mL (6)

ELIGIBILITY:
Inclusion Criteria:

* Male Patients with pathologically proven prostate cancer who will be referred to nuclear medicine unit to perform F18 PSMA for different indications

Exclusion Criteria:

* Undifferentiated prostate cancer.
* Studies with motion artifacts, or those in which patient can't stay stable or calm during acquisition.
* Severely ill patients that hinder imaging.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — male patients with prostate cancer
Study Population: This study will recruit patients with proven prostate cancer who will be referred to the nuclear medicine unit to perform F18-PSMA PET/CT study for initial staging, restaging, evaluation of biochemical recurrence, or follow up
Sampling Method: Non-Probability Sample
Enrollment: 59 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
To correlate between PSA Levels and F-18 PSMA PET/CT Scan findings | baseline
  correlation between PSA Levels and F-18 PSMA PET/CT findings qualitatively & quantitively interpreted by 2 nuclear medicine physicians.
  the Gleason score and findings of anatomical imaging (CT, MRI, ultrasound), will be obtained and compared/correlated with the PSMA expression/volumetric parameters as maximum standardized uptake value (SUV)

SECONDARY OUTCOMES:
To evaluate the impact of PET/CT findings on the patient management | one year
  determine dependency of PSA level in patient management in initial staging or biochemical recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Nadia M Moustafa, PhD degree, Study Director — Assiut University; Aalaa W Hussein, master, Principal Investigator — Assiut University; Mohamed A Mekkawy, PhD degree, Study Chair — Assiut University; Nahla M mahmoud, PhD degree, Study Director — Assiut University
Locations (1):
- Assiut university hospital, Asyut, Egypt

REFERENCES:
- [Background] Tsechelidis I, Vrachimis A. PSMA PET in Imaging Prostate Cancer. Front Oncol. 2022 Jan 28;12:831429. doi: 10.3389/fonc.2022.831429. eCollection 2022. PMID 35155262
- [Background] Liu X, Wang Q, Zhang B, Jiang T, Zeng W. Diagnostic accuracy of 18F-PSMA-1007 PET/CT for prostate cancer in primary staging and biochemical recurrence with different serum PSA levels: A systematic review and meta-analysis. Hell J Nucl Med. 2022 Jan-Apr;25(1):88-102. doi: 10.1967/s002449912438. Epub 2022 Apr 8. PMID 35388806
- [Background] Xu XS, Ryan CJ, Stuyckens K, Smith MR, Saad F, Griffin TW, Park YC, Yu MK, Vermeulen A, Poggesi I, Nandy P. Correlation between Prostate-Specific Antigen Kinetics and Overall Survival in Abiraterone Acetate-Treated Castration-Resistant Prostate Cancer Patients. Clin Cancer Res. 2015 Jul 15;21(14):3170-7. doi: 10.1158/1078-0432.CCR-14-1549. Epub 2015 Mar 31. PMID 25829400
- [Background] Liu X, Jiang T, Gao C, Liu H, Sun Y, Zou Q, Tang R, Zeng W. Detection rate of fluorine-18 prostate-specific membrane antigen-1007 PET/CT for prostate cancer in primary staging and biochemical recurrence with different serum PSA levels: A systematic review and meta-analysis. Front Oncol. 2022 Jul 22;12:911146. doi: 10.3389/fonc.2022.911146. eCollection 2022. PMID 35936732
- [Background] Awenat S, Piccardo A, Carvoeiras P, Signore G, Giovanella L, Prior JO, Treglia G. Diagnostic Role of 18F-PSMA-1007 PET/CT in Prostate Cancer Staging: A Systematic Review. Diagnostics (Basel). 2021 Mar 19;11(3):552. doi: 10.3390/diagnostics11030552. PMID 33808825
- [Result] Tang DG. Understanding and targeting prostate cancer cell heterogeneity and plasticity. Semin Cancer Biol. 2022 Jul;82:68-93. doi: 10.1016/j.semcancer.2021.11.001. Epub 2021 Nov 26. PMID 34844845